CLINICAL TRIAL: NCT06505278
Title: The Impact of Circadian Rhythm-Based Medication Timing Adjustment on the Efficacy and Safety of Novel Hormonal Therapy
Brief Title: The Impact of Medication Timing Adjustment on the Effect of Novel Hormonal Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonghong Li, Chief Physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-183
Record Dates: First submitted 2024-06-23; First posted 2024-07-17 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Circadian Rhythm; Metastatic Hormone-Sensitive Prostate Cancer; Medication Timing; Novel Hormonal Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Night medication group (Experimental): Participants receive Abiraterone plus prednisone/Enzalutamide/Apalutamide/Rezvilutamide between 10:00 pm and 12:00 pm.
  Interventions: Drug: Receive Abiraterone plus prednisone/Enzalutamide/Apalutamide/Rezvilutamide in the evening
- Daytime medication group (No Intervention): Participants receive Abiraterone plus prednisone/Enzalutamide/Apalutamide/Rezvilutamide between 7:00 am and 9:00 am.

INTERVENTIONS:
Drug: Receive Abiraterone plus prednisone/Enzalutamide/Apalutamide/Rezvilutamide in the evening — Participants receive Abiraterone plus prednisone/Enzalutamide/Apalutamide/Rezvilutamide between 10:00 pm and 12:00 pm in the evening.
  Arms: Night medication group

SUMMARY:
The purpose of this study is to assess the impact of medication timing adjustment on the effect of novel hormonal therapy (NHT) agents in patients with metastatic hormone-sensitive prostate cancer (mHSPC). The half of the patients will receive NHT agents in the morning, and the other half will receive NHT agents in the evening.

DETAILED DESCRIPTION:
Metastatic hormone-sensitive prostate cancer (mHSPC) can be treated with androgen deprivation therapy (ADT) plus novel hormonal therapy (NHT) agents such as abiraterone, enzalutamide and apalutamide. However, after a period of treatment, patients inevitably develop resistance to hormonal therapy, progressing to metastatic castration-resistant prostate cancer (mCRPC). Once resistance occurs, treatment options are limited and the prognosis is poor. Therefore, enhancing the efficacy of hormonal therapy and delaying the onset of resistance is currently a focal point of research in advanced prostate cancer.

Androgens are a fundamental basis for the growth, proliferation, and metastasis of prostate cancer cells, exhibiting significant circadian rhythms in their synthesis and secretion. The synthesis of androgens and their products such as androstenedione (A4) and testosterone (T) accelerates in the early morning, peaks around 8:00 AM, then declines, reaching a nadir around 8:00 PM. NHT agents, such as abiraterone, primarily inhibit the synthesis of androgens by blocking the CYP17A1 enzyme, thereby aiming to suppress tumor growth. However, abiraterone is currently administered mainly on an empty stomach in the morning, when androgen and its metabolites have already peaked and been released into the bloodstream. Hence, inhibiting androgen synthesis at this time may not yield optimal effects.

Chronotherapy refers to the administration of therapy in alignment with the circadian rhythms of the patient, tumor, and drug to enhance therapeutic efficacy and reduce adverse reactions. In certain malignancies, research has been conducted to adjust the timing of drug administration based on these circadian characteristics, resulting in improved efficacy and reduced adverse reactions compared to traditional dosing schedules.

However, no study has explored the impact of different timing of NHT agents administration on the therapeutic efficacy and safety currently.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily participate in the study and have signed a written informed consent form (ICF);
* Male patients aged 18 to 75 years (inclusive) at the time of signing the ICF;
* Histologically or cytologically confirmed prostate cancer, without prior novel hormonal therapy (NHT) or chemotherapy;
* Assessed as having metastatic hormone-sensitive prostate cancer (mHSPC), defined as: histologically or cytologically confirmed prostate cancer with distant metastases (beyond regional lymph nodes) detected by bone scan, MRI, CT, PET/CT, or pathological examination, and who have not received hormonal therapy or chemotherapy;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1;
* Normal routine blood count and liver and kidney functions, expected to tolerate treatment for mHSPC;
* Expected survival period ≥ 12 weeks.
* Agreement to sign the ICF.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria;
* Patients currently receiving other systemic anticancer treatments (such as chemotherapy and/or immunotherapy);
* Patients who have undergone organ transplantation within the past three months;
* Patients with active, known, or suspected autoimmune diseases; or those testing positive for hepatitis B virus, hepatitis C virus, or HIV indicating acute or chronic infection;
* Patients with severe life-threatening diseases;
* Patients who have not signed the ICF;
* Other conditions deemed by the researchers to make the patient unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PSA response rate defiend as the proportion of participants whose prostate specific antigen (PSA) decreases by more than 90% from baseline after three months of treatment | Baseline and Week 12
  PSA is a critical indicator for assessing the efficacy of prostate cancer treatment; typically, a lower PSA value suggests better therapeutic outcomes. A second PSA measurement is confirmed after 3 weeks from week 12.

SECONDARY OUTCOMES:
Circulating tumor cell (CTC) clearance rate defiend as the proportion testing negative for circulating tumor cell (CTC) at week 12 in patients with a baseline CTC count of ≥1 | Baseline and Week 12
  CTC are tumor cells that enter the bloodstream and are associated with the metastasis of tumors. Typically, a lower CTC count is indicative of better therapeutic efficacy.
Clinical benefit rate (CBR) defiend as the proportion of patients comfirming partial response (PR), complete response (CR), or stable disease (SD). | Through study completion, an average of 18 months
  Clinical benefit refers to participants achieving PR, CR, or SD.
Objective response rate (ORR) defiend as the proportion of participants confirming partial response (PR) or complete response (CR) | Through study completion, an average of 18 months
  Objective response refers to participants achieving PR or CR, which would be confirmed 4 weeks later.
Duration of relief defiend from the first assessment of complete response (CR) or partial response (PR) until the detection of disease progression (PD) | From CR or PR to PD, up to 18 months
  Duration of relief represents the length of time the tumor remains reduced under this treatment regimen.
Time to achieve objective relief defiend from randomization until achieving complete response (CR) or partial response (PR). | From start of treatment to CR or PR, up to 18 months
  Time to achieve objective relief is an important indicator of therapeutic efficacy.
Time to PSA progression defiend the time from detection of PSA nadir to PSA progression | From start of treatment to PSA progression, up to 18 months
  PSA progression refers to PSA>1ng/ml, with at least a one-week interval between PSA measurement and two consecutive increases of>50% compared to the baseline value.
Radiographic progression-free survival (rPFS) defiend from randomization until radiographic progression according to RECIST 1.1 criteria | From start of treatment to radiographic progression, up to 18 months
  rPFS refers to the time from randomization to radiographic progression defined as tumor progression assessed by CT, MRI, or ECT according to RECIST 1.1 criteria, which is an important indicator for treatment efficacy.
Overall survival defined from randomization until death from any cause. | From start of treatment to death from any cause, up to 18 months
  Time to death refers to the time from randomization to death from any cause, which is a crucial indicator for treatment efficacy.
Treatment emerged adverse event (TEAE) | Throughout the entire study period，an average of 18 months
  Treatment emerged adverse event would be assessed by NCI-CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghong Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Mottet N, Cornford P, Vanden Bergh RCN, et al. EAU-EANM-ESTRO-ESUR-ISUP_SIOG guidelines on prostate cancer. (2023).
- [Background] Schaeffer EM, Srinivas S, Adra N, An Y, Barocas D, Bitting R, Bryce A, Chapin B, Cheng HH, D'Amico AV, Desai N, Dorff T, Eastham JA, Farrington TA, Gao X, Gupta S, Guzzo T, Ippolito JE, Kuettel MR, Lang JM, Lotan T, McKay RR, Morgan T, Netto G, Pow-Sang JM, Reiter R, Roach M, Robin T, Rosenfeld S, Shabsigh A, Spratt D, Teply BA, Tward J, Valicenti R, Wong JK, Shead DA, Snedeker J, Freedman-Cass DA. Prostate Cancer, Version 4.2023, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2023 Oct;21(10):1067-1096. doi: 10.6004/jnccn.2023.0050. PMID 37856213
- [Background] Ryan CJ, Smith MR, Fizazi K, Saad F, Mulders PF, Sternberg CN, Miller K, Logothetis CJ, Shore ND, Small EJ, Carles J, Flaig TW, Taplin ME, Higano CS, de Souza P, de Bono JS, Griffin TW, De Porre P, Yu MK, Park YC, Li J, Kheoh T, Naini V, Molina A, Rathkopf DE; COU-AA-302 Investigators. Abiraterone acetate plus prednisone versus placebo plus prednisone in chemotherapy-naive men with metastatic castration-resistant prostate cancer (COU-AA-302): final overall survival analysis of a randomised, double-blind, placebo-controlled phase 3 study. Lancet Oncol. 2015 Feb;16(2):152-60. doi: 10.1016/S1470-2045(14)71205-7. Epub 2015 Jan 16. PMID 25601341
- [Background] Beer TM, Armstrong AJ, Rathkopf DE, Loriot Y, Sternberg CN, Higano CS, Iversen P, Bhattacharya S, Carles J, Chowdhury S, Davis ID, de Bono JS, Evans CP, Fizazi K, Joshua AM, Kim CS, Kimura G, Mainwaring P, Mansbach H, Miller K, Noonberg SB, Perabo F, Phung D, Saad F, Scher HI, Taplin ME, Venner PM, Tombal B; PREVAIL Investigators. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Jul 31;371(5):424-33. doi: 10.1056/NEJMoa1405095. Epub 2014 Jun 1. PMID 24881730
- [Background] Zhou T, Zeng SX, Ye DW, Wei Q, Zhang X, Huang YR, Ye ZQ, Yang Y, Zhang W, Tian Y, Zhou FJ, Jie J, Chen SP, Sun Y, Xie LP, Yao X, Na YQ, Sun YH. A multicenter, randomized clinical trial comparing the three-weekly docetaxel regimen plus prednisone versus mitoxantone plus prednisone for Chinese patients with metastatic castration refractory prostate cancer. PLoS One. 2015 Jan 27;10(1):e0117002. doi: 10.1371/journal.pone.0117002. eCollection 2015. PMID 25625938
- [Background] Ozturk N, Ozturk D, Kavakli IH, Okyar A. Molecular Aspects of Circadian Pharmacology and Relevance for Cancer Chronotherapy. Int J Mol Sci. 2017 Oct 17;18(10):2168. doi: 10.3390/ijms18102168. PMID 29039812
- [Background] Patke A, Young MW, Axelrod S. Molecular mechanisms and physiological importance of circadian rhythms. Nat Rev Mol Cell Biol. 2020 Feb;21(2):67-84. doi: 10.1038/s41580-019-0179-2. Epub 2019 Nov 25. PMID 31768006
- [Background] Rosenwasser AM, Turek FW. Neurobiology of Circadian Rhythm Regulation. Sleep Med Clin. 2015 Dec;10(4):403-12. doi: 10.1016/j.jsmc.2015.08.003. Epub 2015 Sep 11. PMID 26568118
- [Background] Hastings MH, Maywood ES, Brancaccio M. Generation of circadian rhythms in the suprachiasmatic nucleus. Nat Rev Neurosci. 2018 Aug;19(8):453-469. doi: 10.1038/s41583-018-0026-z. PMID 29934559
- [Background] Turcu AF, Zhao L, Chen X, Yang R, Rege J, Rainey WE, Veldhuis JD, Auchus RJ. Circadian rhythms of 11-oxygenated C19 steroids and ∆5-steroid sulfates in healthy men. Eur J Endocrinol. 2021 Aug 27;185(4):K1-K6. doi: 10.1530/EJE-21-0348. PMID 34324429
- [Background] Rivard GE, Infante-Rivard C, Hoyoux C, Champagne J. Maintenance chemotherapy for childhood acute lymphoblastic leukaemia: better in the evening. Lancet. 1985 Dec 7;2(8467):1264-6. doi: 10.1016/s0140-6736(85)91551-x. PMID 2866334
- [Background] Rivard GE, Infante-Rivard C, Dresse MF, Leclerc JM, Champagne J. Circadian time-dependent response of childhood lymphoblastic leukemia to chemotherapy: a long-term follow-up study of survival. Chronobiol Int. 1993 Jun;10(3):201-4. doi: 10.3109/07420529309073888. PMID 8319318
- [Background] Qian DC, Kleber T, Brammer B, Xu KM, Switchenko JM, Janopaul-Naylor JR, Zhong J, Yushak ML, Harvey RD, Paulos CM, Lawson DH, Khan MK, Kudchadkar RR, Buchwald ZS. Effect of immunotherapy time-of-day infusion on overall survival among patients with advanced melanoma in the USA (MEMOIR): a propensity score-matched analysis of a single-centre, longitudinal study. Lancet Oncol. 2021 Dec;22(12):1777-1786. doi: 10.1016/S1470-2045(21)00546-5. Epub 2021 Nov 12. PMID 34780711
- [Background] Ryan CJ, Smith MR, Fong L, Rosenberg JE, Kantoff P, Raynaud F, Martins V, Lee G, Kheoh T, Kim J, Molina A, Small EJ. Phase I clinical trial of the CYP17 inhibitor abiraterone acetate demonstrating clinical activity in patients with castration-resistant prostate cancer who received prior ketoconazole therapy. J Clin Oncol. 2010 Mar 20;28(9):1481-8. doi: 10.1200/JCO.2009.24.1281. Epub 2010 Feb 16. PMID 20159824
- [Background] Hong JH. Pharmacokinetic/pharmacodynamic drug evaluation of enzalutamide for treating prostate cancer. Expert Opin Drug Metab Toxicol. 2018 Mar;14(3):361-369. doi: 10.1080/17425255.2018.1440288. Epub 2018 Feb 13. PMID 29431540